CLINICAL TRIAL: NCT06266546
Title: Prophylactic Endobronchial Tranexamic Acid to Reduce Bleeding in Transbronchial Cryobiopsy
Acronym: CRYOTXA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Youssef Yammine (Other)
Responsible Party: Sponsor-Investigator, Youssef Yammine, Principal Investigator, Ascension Via Christi Hospitals Wichita, Inc.
Organization: Ascension Via Christi Hospitals Wichita, Inc. (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRYOTXA
Record Dates: First submitted 2024-01-10; First posted 2024-02-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hemorrhage Lung; Endobronchial Mass
Keywords: Transbronchial biopsy; Tranexamic Acid (TXA); Hemorrhage; Prophylaxis
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, single-arm, non-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Prophylactic TXA arm
  Interventions: Drug: Tranexamic acid
- Control (No Intervention): Data collected retrospectively from patients undergoing the same procedure one year prior to the study initiation

INTERVENTIONS:
Drug: Tranexamic acid — Prophylactic tranexamic acid will be instilled via endobronchial route in all patients undergoing transbronchial cryobiopsy. The medication will be administered through the bronchoscope one minute prior to the cryobiopsy. 500 mg of TXA diluted in 10 ml of saline and the procedure would be carried out as usual.
  Arms: Intervention

SUMMARY:
Transbronchial cryobiopsies are common procedures used to obtain tissue samples from airways for diagnostic purposes. While these procedures are safe, there is a risk of bleeding from the biopsy site. We are conducting a research study to assess the safety and effectiveness of using tranexamic acid prior to undergoing a transbronchial cryobiopsy.

DETAILED DESCRIPTION:
Prophylactic tranexamic acid will be instilled via endobronchial route in all patients undergoing transbronchial cryobiopsy. The medication will be administered through the bronchoscope one minute prior to the cryobiopsy. 500 mg of TXA diluted in 10 ml of saline and the procedure would be carried out as usual.

The study will be a prospective, single-arm, non-randomized trial Location: Ascension Via Christi Saint Francis. Medication: Tranexamic acid 500 milligrams per 5 mL ampule (Baxter, NDC 43066-008-01) mixed with 10 mL normal saline.

Patients: A total of 100 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Signed informed consent
* Receiving a transbronchial cryobiopsy

Exclusion Criteria:

* Age below 18
* Pregnancy
* Bleeding diathesis (INR >1.5 or known hematological problems)
* Subarachnoid hemorrhage
* Any active bleeding (any site)
* Decompensated liver disease
* Active intravascular clotting
* Prior VTE
* On oral contraceptive therapy
* Platelet count less than 50,000
* Use of antiplatelet medication other than low-dose aspirin within 5 days of procedure
* Use of therapeutic anticoagulation within the last 24 hrs
* Known severe pulmonary hypertension (pulmonary artery systolic pressure > 60 mmHg)
* Chronic renal failure (estimated GFR below 30 mL/min)
* Allergy or hypersensitivity to tranexamic acid or any of its ingredients
* Prisoners
* Comfort care planned or initiated within 72 hours of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Major Hemorrhage | up to 2 hours post procedure
  Ordinal scale of less severe to most severe
  1. No hemorrhage 2. Minor hemorrhage 3. Intermediate hemorrhage 4. Major hemorrhage

SECONDARY OUTCOMES:
Early termination of the procedure due to bleeding | up to 2 hours post procedure
Rate of intermediate hemorrhage | up to 2 hours post procedure
Rate of minor hemorrhage | up to 2 hours post procedure
Inadequate tissue sampling due to bleeding | up to 2 hours post procedure
  y/n
Graded use of other measures to control bleeding (not prophylactic) | up to 2 hours post procedure
  In order of escalating interventions (severity): use of iced saline, epinephrine, mainstem intubation, embolization
Unplanned hospital admission for bleeding complications | 2 hours post procedure uo to 30 days post procedure
  hospital readmission
Acute cardiovascular side effects | up to 30 days post procedure
  thrombosis events
All cause 28 day mortality | up to 28 days post procedure
  morality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Via Christi, Wichita, Kansas, United States

REFERENCES:
- [Background] Babiak A, Hetzel J, Krishna G, Fritz P, Moeller P, Balli T, Hetzel M. Transbronchial cryobiopsy: a new tool for lung biopsies. Respiration. 2009;78(2):203-8. doi: 10.1159/000203987. Epub 2009 Feb 21. PMID 19246874
- [Background] Hetzel J, Eberhardt R, Petermann C, Gesierich W, Darwiche K, Hagmeyer L, Muche R, Kreuter M, Lewis R, Ehab A, Boeckeler M, Haentschel M. Bleeding risk of transbronchial cryobiopsy compared to transbronchial forceps biopsy in interstitial lung disease - a prospective, randomized, multicentre cross-over trial. Respir Res. 2019 Jul 5;20(1):140. doi: 10.1186/s12931-019-1091-1. PMID 31277659
- [Background] Bendstrup E, Kronborg-White S, Poletti V, Folkersen B, Voldby N, Rasmussen TR. Careful Planning Reduces Cryobiopsy Complications. Ann Am Thorac Soc. 2017 Jul;14(7):1229. doi: 10.1513/AnnalsATS.201703-196LE. No abstract available. PMID 28665702
- [Background] Cai J, Ribkoff J, Olson S, Raghunathan V, Al-Samkari H, DeLoughery TG, Shatzel JJ. The many roles of tranexamic acid: An overview of the clinical indications for TXA in medical and surgical patients. Eur J Haematol. 2020 Feb;104(2):79-87. doi: 10.1111/ejh.13348. Epub 2019 Dec 16. PMID 31729076
- [Background] Zhou GW, Zhang W, Dong YC, Huang HD, Hu C, Sun J, Jin F, Gu Y, Li Q, Li S. Flexible bronchoscopy-induced massive bleeding: A 12-year multicentre retrospective cohort study. Respirology. 2016 Jul;21(5):927-31. doi: 10.1111/resp.12784. Epub 2016 Apr 8. PMID 27061330
- [Background] Pabinger I, Fries D, Schochl H, Streif W, Toller W. Tranexamic acid for treatment and prophylaxis of bleeding and hyperfibrinolysis. Wien Klin Wochenschr. 2017 May;129(9-10):303-316. doi: 10.1007/s00508-017-1194-y. Epub 2017 Apr 21. PMID 28432428
- [Background] Marquez-Martin E, Vergara DG, Martin-Juan J, Flacon AR, Lopez-Campos JL, Rodriguez-Panadero F. Endobronchial administration of tranexamic Acid for controlling pulmonary bleeding: a pilot study. J Bronchology Interv Pulmonol. 2010 Apr;17(2):122-5. doi: 10.1097/LBR.0b013e3181dc8c17. PMID 23168726
- [Background] Kuint R, Levy L, Cohen Goichman P, Huszti E, Abu Rmeileh A, Shriki O, Abutbul A, Fridlender ZG, Berkman N. Prophylactic use of tranexamic acid for prevention of bleeding during transbronchial lung biopsies - A randomized, double-blind, placebo-controlled trial. Respir Med. 2020 Nov;173:106162. doi: 10.1016/j.rmed.2020.106162. Epub 2020 Sep 21. PMID 32979620